CLINICAL TRIAL: NCT06133322
Title: Blood Pressure Lowering Strategies to Eliminate Hypertension Disparities
Brief Title: Blood Pressure Lowering Strategies to Eliminate Hypertension Disparities (BLESSED)
Acronym: BLESSED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Jiang He, MD, PhD, Director Tulane University Translational Science Institute, Tulane University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-1081-SPHTM; R01MD018193 (NIH)
Record Dates: First submitted 2023-11-01; First posted 2023-11-15 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2024-05

CONDITIONS: Hypertension
Keywords: church-based; Black; African American; Community-based Intervention; health disparities; cardiovascular disease prevention
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Cluster randomization of 42 churches in New Orleans, Louisiana to 2 arms
Who Masked: Outcomes Assessor
Masking Description: Clinical research coordinators and laboratory technicians who assess health-related outcomes will be blinded to intervention assignment. Study physicians who review serious adverse events and unanticipated problems will also be blinded to intervention assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Community health worker-led implementation strategy (Experimental): CHW-led church-based multifaceted implementation strategy: CHWs will conduct individualized health coaching and healthcare navigation, organize church-based health promotion programs (e.g., nutrition education and exercise sessions), and train and assist the study participants in self-monitoring of BP. Nurse practitioners will see study participants at church settings, and community pharmacies will deliver antihypertensive medications to patients' homes.
  Interventions: Behavioral: Behavioral: Evidence-based interventions recommended by the 2017 ACC/AHA hypertension clinical guideline
- Group-based Education Strategy (Experimental): The investigator team will work with church leadership and wellness coordinators to organize group-based education sessions. Health education will be delivered by local primary care providers, dieticians, and health educators. Contact information for primary care providers and information on self-monitoring of BP will also be given at group sessions.
  Interventions: Behavioral: Behavioral: Evidence-based interventions recommended by the 2017 ACC/AHA hypertension clinical guideline

INTERVENTIONS:
Behavioral: Behavioral: Evidence-based interventions recommended by the 2017 ACC/AHA hypertension clinical guideline — The recommended evidence-based interventions include therapeutic lifestyle change and medical treatment of hypertension

SUMMARY:
The burden of hypertension and related cardiovascular diseases, stroke, and end-stage kidney disease is disproportionately high in Black populations, especially in the South. The Blood Pressure Lowering Strategies to Eliminate Hypertension Disparities (BLESSED) cluster randomized trial aims to test the effectiveness, implementation, and sustainability of a community health worker (CHW)-led multifaceted intervention compared to enhanced usual care for hypertension control in Black communities. In the BLESSED trial, the investigators plan to recruit 1,176 adults with hypertension (approximately 28 per church) from 42 predominantly Black churches in the Greater New Orleans area. The multifaceted intervention will last for 18 months, followed by a post-intervention follow-up visit at 24 months. The BLESSED trial aims to generate evidence regarding the effectiveness, implementation, and sustainability of this CHW-led church-based multifaceted intervention in eliminating hypertension disparities in the United States (US) general population.

DETAILED DESCRIPTION:
Louisiana residents, especially African Americans, bear a disproportionately high burden of hypertension and cardiovascular disease (CVD). In the Blood Pressure Lowering Strategies to Eliminate Hypertension Disparities (BLESSED) cluster randomized trial, the investigators will compare the impact of two implementation strategies - a CHW-led multifaceted strategy and a group-based education strategy - for delivering interventions recommended by the 2017 American College of Cardiology (ACC) and the American Heart Association (AHA) hypertension clinical guidelines on implementation and clinical effectiveness outcomes in predominantly Black community members over 18 months. The BLESSED study utilizes an effectiveness-implementation hybrid design to: (1). test the effectiveness of a CHW-led church-based multifaceted implementation strategy for reducing estimated CVD risk over 18 months among African American church community members at high risk for CVD, and (2). assess the implementation outcomes (acceptability, adaptation, adoption, feasibility, fidelity, penetrance, cost-effectiveness, and sustainability) simultaneously. The Exploration, Preparation, Implementation, Sustainment (EPIS) framework has guided the development and evaluation of the multifaceted implementation strategy, which includes CHW-led health coaching on lifestyle changes and medication adherence; healthcare delivery in community; church-based exercise and weight loss programs; self-monitoring of blood pressure (BP); and provider education and engagement. The CHW-led church-based intervention will provide strong social support and tackle multiple social determinants of CVD disparities. The primary clinical effectiveness outcome is the difference in mean change of systolic blood pressure (SBP) from baseline to 18 months between intervention and control groups. The primary implementation outcome is a fidelity summary score for key implementation strategy components to the CHW-led church-based multifaceted implementation strategy assessed at the participant levels. This study has 90% statistical power to detect group differences in mean SBP change of 5.8 mm Hg over 18 months using a 2-sided significance level of 0.05. The investigators will recruit 1,176 participants (28 per church) who are aged ≥18 years with systolic blood pressure ≥130 mmHg or diastolic blood pressure ≥80 mm Hg, and randomly assign 21 churches to intervention and 21 to control; the investigators will implement the multifaceted intervention program; the investigators will follow-up participants and collect data on effectiveness and implementation outcomes at 6, 12, and 18 months; the investigators will evaluate the sustainability of the intervention at 6 months post-intervention; and the investigators will perform intention-to-treat analyses and disseminate and scale-up the proven-effective implementation strategy. The proposed study will generate evidence on the effectiveness, implementation, and sustainability of the multifaceted intervention aimed at eliminating CVD disparities in African American populations in the US.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged ≥18 years
2. Community members associated with the participating churches (church members and their families and friends)
3. Systolic blood pressure ≥130 mmHg or diastolic blood pressure ≥80 mm Hg
4. Willing and able to participate in the intervention.
5. Willing and able to sign written informed consent.

Exclusion Criteria:

1. Prior hospitalization in the last 3 months for chronic heart failure or heart attack
2. Current diagnosis of cancer requiring chemotherapy or radiation therapy
3. Stage-5 chronic kidney disease requiring chronic dialysis or transplant
4. Pregnant or planning to become pregnant in the next 18 months
5. Planning to move out of the Greater New Orleans area during the next year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1176 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Difference in mean change of systolic blood pressure | Measured from baseline to 18 months
  Difference in mean change of systolic blood pressure from baseline to 18 months between intervention and control groups
Implementation fidelity summary score | Measured at 6, 12, and 18 months
  The fidelity summary score is composed of the following key implementation strategy components: proportion of assigned health education sessions attended in all participants, proportion of assigned discussion sessions attended in all participants, proportion of recommended minutes of physical activity completed in all participants, proportion of days per week that fruits/vegetables are eaten as recommended in all participants, proportion of recommended home blood pressure (BP) monitoring completed in patients with hypertension, proportion of required provider visits attended in all patients, and proportion of antihypertensive medications taken in patients with hypertension. The score ranged from zero to six with a higher score indicates greater fidelity.

SECONDARY OUTCOMES:
Difference in the proportion of patients with controlled BP between intervention and control groups | Measured from baseline to 18 months
  Difference in the proportion of patients with controlled BP (<130/80 mm Hg) between intervention and control groups at 18 months
Difference in mean change of diastolic BP | Measured from baseline to 18 months
  Difference in mean change of diastolic BP (DBP) from baseline to 18 months between intervention and control groups
Side effects of medications and adverse events | Measured from baseline to 18 months
  Change in side effects of medications and adverse events from baseline to 18 months
Cost-effectiveness | Measured from baseline to 18 months
  Cost-effectiveness assessed as incremental direct costs per additional percentage of hypertension control
Acceptability | Measured from baseline to 18 months
  Percentage of participants, community health worker, providers, and church administrators who reply that the intervention is acceptable (satisfactory). Measured by survey.
Adoption (Churches) | Measured from baseline to 18 months
  % of churches adopting the intervention program
Adoption (Providers) | Measured from baseline to 18 months
  % of invited providers attending training sessions
Appropriateness | Measured from baseline to 18 months
  Percentage of participants, community health workers, providers, and church administrators who reply that the intervention is appropriate (good perceived fit). The outcome will be measured by survey question.
Feasibility to participant, community health worker, provider and churches | Measured from baseline to 18 months
  Percentage of participants, community health worker, providers, and church administrators who reply that the intervention is feasible (actual fit, suitability). Measured by survey and study administrative data.
Exercise Session Fidelity (community health worker-led strategy group) | Measured at 6, 12, and 18 months
  Percentage of exercise sessions organized. Measured by study administrative data.
Fidelity of Group Health Education Session | Measured at 6, 12, and 18 months
  Percentage of group health education sessions conducted out of health educated sessions planned per study protocol.
Nutrition Education Session Fidelity (community health worker-led strategy group) | Measured at 6, 12, and 18 months
  Percentage of nutrition education sessions organized. Measured by study administrative data.
Health Care Appointment Fidelity (community health worker-led strategy group) | Measured at 6, 12, and 18 months
  Percentage of health care visit appointments made. Measured by study administrative data.
Percentage of enrolled participants receiving assigned intervention. Measured by study administrative data. Reach (Participants) | Measured at baseline, 6, 12, and 18 months
  Percentage of enrolled participants receiving assigned intervention. Measured by study administrative data.
Reach (Participants) | Measured at baseline
  The percentage of eligible/screened/contacted participants enrolled. Measured by study data, administrative data.
Penetrance (Participants) | Measured at baseline, 6, 12, and 18 months
  Percentage of enrolled participants receiving assigned intervention. Measured by intervention monitoring data.
Penetrance (Providers) | Measured at baseline, 6, 12, and 18 months
  Percentage of trained providers delivering protocol-based care. Measured by intervention monitoring data.
Penetrance (educators) | Measured at baseline, 6, 12, and 18 months
  Percentage of trained CHWs or providers and health educators delivering health coaching. Measured by intervention monitoring data.
Sustainability (Churches) | Measured at baseline, 6, 12, and 18 months
  Percentage of churches continuing the intervention program and individual components. Measured by 6-month post-intervention survey.
Sustainability (Participants) | Measured at 24 months
  Percentage of participants maintaining ideal cardiovascular health metrics, healthy lifestyle components, and adherence to medications. Measured by 6-month post-intervention survey and examination.
Sustainability Effectiveness Outcome: Differences in mean change of SBP and DBP | Measured at baseline and 24 months
  Differences in mean change of SBP and DBP from baseline to 24 months (6 months post-intervention) between intervention and control groups
Sustainability Effectiveness Outcome: Difference in the proportion of patients with controlled BP | Measured at baseline and 24 months
  Difference in the proportion of patients with controlled BP (<130/80 mm Hg) between intervention and control groups at 24 months.
Sustainability of Fidelity | Measured at 24 months
  A fidelity summary score for key implementation strategy components at 6 months post-intervention (24 months overall). The fidelity summary score is composed of the following key implementation strategy components: proportion of assigned health education sessions attended in all participants, proportion of assigned discussion sessions attended in all participants, proportion of recommended minutes of physical activity completed in all participants, proportion of days per week that fruits/vegetables are eaten as recommended in all participants, proportion of recommended home BP monitoring completed in patients with hypertension, proportion of required provider visits attended in all patients, and proportion of antihypertensive medications taken in patients with hypertension. Fidelity score ranges from zero to six with a higher score indicates greater fidelity.

OTHER OUTCOMES:
Change in quality of life | Measured from baseline to 18 months
  The difference in QoL between the two arms over 18 months. QoL will be assessed using the SF-12 questionnaire. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- Tulane University, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
The study data sharing plan will comply with all NIH policies for data sharing. Data sharing will be executed through the centralized NIH data repository and will be implemented in a timely manner. The study data, including data from baseline and follow-up visits, will be prepared for transmission to the NHLBI data repository - the Biologic Specimen and Data Repository Information Coordinating Center (BioLINCC). The datasets will be submitted to the NHLBI no later than three years after the end of the final participant follow-up or two years after the main paper of the trial has been published, whichever comes first. The NHLBI will review the submitted data prior to release. These data will be free of identifiers that allow identification of individual research participants either directly or through "deductive disclosure." In addition, the investigators will offer, through a publicly accessible website, opportunities for outside investigators to collaborate using complete study data.
Supporting Information: Study Protocol, SAP
Time Frame: No later than three years after the end of the final participant follow-up or two years after the main paper of the trial has been published, whichever comes first

REFERENCES:
- [Background] Maroney K, Laurent J, Alvarado F, Gabor A, Bell C, Ferdinand K, He J, Mills KT. Systematic review and meta-analysis of church-based interventions to improve cardiovascular disease risk factors. Am J Med Sci. 2023 Sep;366(3):199-208. doi: 10.1016/j.amjms.2023.05.010. Epub 2023 May 25. PMID 37244637
- [Background] He J, Bundy JD, Geng S, Tian L, He H, Li X, Ferdinand KC, Anderson AH, Dorans KS, Vasan RS, Mills KT, Chen J. Social, Behavioral, and Metabolic Risk Factors and Racial Disparities in Cardiovascular Disease Mortality in U.S. Adults : An Observational Study. Ann Intern Med. 2023 Sep;176(9):1200-1208. doi: 10.7326/M23-0507. Epub 2023 Aug 15. PMID 37579311
- [Background] Bundy JD, Mills KT, He H, LaVeist TA, Ferdinand KC, Chen J, He J. Social determinants of health and premature death among adults in the USA from 1999 to 2018: a national cohort study. Lancet Public Health. 2023 Jun;8(6):e422-e431. doi: 10.1016/S2468-2667(23)00081-6. PMID 37244672